CLINICAL TRIAL: NCT01329913
Title: A Multiple Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of MK-6325 in Hepatitis C Infected Male and Female Patients
Brief Title: Safety, Pharmacokinetics, and Pharmacodynamics of MK-6325 in Hepatitis C Virus (HCV) Infections (MK-6325-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6325-003; 2010-023687-40 (EudraCT Number)
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — MK-6325

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- GT1-HCV 200 mg (Experimental)
  Interventions: Drug: MK-6325; Drug: Placebo to MK-6325
- GT1-HCV 400 mg (Experimental)
  Interventions: Drug: MK-6325; Drug: Placebo to MK-6325
- GTI-HCV 800 mg (Experimental)
  Interventions: Drug: MK-6325; Drug: Placebo to MK-6325
- GT3-HCV 200 mg (Experimental)
  Interventions: Drug: MK-6325; Drug: Placebo to MK-6325
- GT3-HCV 400 mg (Experimental)
  Interventions: Drug: MK-6325; Drug: Placebo to MK-6325
- GT3-HCV 800 mg (Experimental)
  Interventions: Drug: MK-6325; Drug: Placebo to MK-6325

INTERVENTIONS:
Drug: MK-6325 — Two 100 mg capsules, orally, once per day for 7 days
  Arms: GT1-HCV 200 mg; GT3-HCV 200 mg
Drug: Placebo to MK-6325 — Two 100 mg capsules, orally, once per day for 7 days
  Arms: GT1-HCV 200 mg; GT3-HCV 200 mg
Drug: MK-6325 — Four 100 mg capsules, orally, once per day for 7 days
  Arms: GT1-HCV 400 mg; GT3-HCV 400 mg
Drug: Placebo to MK-6325 — Four 100 mg capsules, orally, once per day for 7 days
  Arms: GT1-HCV 400 mg; GT3-HCV 400 mg
Drug: MK-6325 — Eight 100 mg capsules, orally, once per day for 7 days
  Arms: GT3-HCV 800 mg; GTI-HCV 800 mg
Drug: Placebo to MK-6325 — Eight 100 mg capsules, orally, once per day for 7 days
  Arms: GT3-HCV 800 mg; GTI-HCV 800 mg

SUMMARY:
This is a 2 part study of the safety, pharmacokinetics and pharmacodynamics of MK-6325 in HCV-infected participants. Part I of the study will be for Genotype (GT) 1 HCV-infected participants who will be randomized to receive either MK-6325 or placebo. If the drug is shown to be safe and efficacious in Part I, Part II will enroll GT 3 HCV-infected participants who will be randomized to receive either MK-6325 or placebo.

ELIGIBILITY:
Inclusion criteria:

* Body mass index (BMI) of 18 to ≤37 kg/m^2.
* Stable health
* No clinically significant abnormality on electrocardiogram (ECG)
* Clinical diagnosis of chronic HCV infection (G1 or G3) for at least 6 months and detectable HCV RNA in peripheral blood.

Exclusion criteria:

* Pregnancy or intention to become pregnant or father a child during the course of the study.
* History of stroke, chronic seizures, major neurological disorder, or uncontrolled clinically significant psychiatric disorder (for example, depression).
* Estimated creatinine clearance of ≤70 mL/min.
* History of clinically significant endocrine, gastrointestinal (except HCV infection), cardiovascular, hematological, immunological, renal, respiratory, or genitourinary abnormalities or diseases whose current condition is considered clinically unstable.
* History of neoplastic disease other than adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix ≥10 years prior to the prestudy (screening) visit with no evidence of recurrence of likelihood of recurrence.
* Positive Hepatitis B surface antigen at the pre-study (screening) visit.
* History of documented HIV infection or positive HIV serology at the pre-study (screening) visit.
* Regular consumption of excessive amounts of alcohol, defined as greater than 2 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day.
* Excessive consumption, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) or coffee, tea, cola, or other caffeinated beverages per day.
* Major surgery, or donation or loss of 1 unit of blood (approximately 500 mL) or participated in another investigational study within 4 weeks prior to the prestudy (screening) visit.
* History of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food.
* Regular use of (including "recreational use") of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 2 months. Exception: marijuana use is permitted at the discretion of the investigator and provided the participant can refrain from its use during the study.
* Evidence or history of chronic hepatitis not caused by HCV including but not limited to non-HCV viral hepatitis, non-alcoholic steatohepatitis (NASH), drug-induced hepatitis, autoimmune hepatitis. Note: Participants with history of acute non-HCV-related hepatitis, which resolved >6 months before study can be enrolled.
* Previous treatment with other HCV protease inhibitors ≤3 months prior to the first dose of study drug.
* Previous exposure to interferon-alpha and/or ribavirin within 3 month prior to the first dose of MK-6325 in the study.
* Clinical or laboratory evidence of advanced or decompensated liver disease; evidence of bridging fibrosis or higher grade fibrosis (Metavir score ≥3) from prior liver biopsy. Note: liver biopsy is not required for entry into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing clinical and laboratory adverse events (AEs) (Parts I and II) | Up to 15 days after last dose of study drug

SECONDARY OUTCOMES:
Viral load reduction in GT1 HCV-infected participants (Part I) | 7 Days
Viral load reduction in GT3 HCV-infected participants (Part II) | 7 Days